CLINICAL TRIAL: NCT05955924
Title: Nicotinamide Chemoprevention for Keratinocyte Carcinoma in Solid Organ Transplant Recipients: a Multicentre, Pragmatic Randomized Trial
Brief Title: Nicotinamide Chemoprevention for Keratinocyte Carcinoma in Solid Organ Transplant Recipients - Pivotal Trial
Acronym: SPRINTR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University Health Network, Toronto (Other); NOW Foods (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPRINTR-pivotal
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Non-melanoma Skin Cancer; Carcinoma, Squamous Cell; Carcinoma, Basal Cell; Keratinocyte Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: Multicentre, parallel group, placebo-controlled, pragmatic randomized trial with 1:1 allocation and a superiority framework
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental): Intervention Drug : Nicotinamide
  Interventions: Drug: Nicotinamide
- Placebo (Placebo Comparator): Intervention: Placebo Oral Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide — Oral nicotinamide (500 mg) twice daily
  Other Names: niacinamide
  Arms: Nicotinamide
Drug: Placebo — Matching placebo capsule twice daily
  Arms: Placebo

SUMMARY:
As patients live longer after receiving an organ transplant, there is a need to reduce the long-term side effects of the drugs used to prevent organ rejection. In particular, long-term use of these drugs increases the risk of skin cancer. Skin cancer is now a leading cause of illness and disfigurement after kidney, liver, heart, and lung transplantation. Given the increased risk and burden of skin cancer in transplant recipients, prevention is critical.

Nicotinamide is a form of Vitamin B3 that has been shown to protect against skin cancer in the general population. However, it is unclear whether nicotinamide is effective among immune-suppressed transplant recipients. Investigators will conduct a clinical trial involving multiple transplant centres in Canada to evaluate whether oral nicotinamide (500 mg twice daily) is effective and safe for preventing skin cancer. Investigators will recruit 396 high-risk adult kidney, liver, heart, and lung transplant patients who have previously had at least one skin cancer. Patients will receive nicotinamide or sham tablets for up to 4 years. The results will inform efforts to improve the long-term health of transplant recipients.

DETAILED DESCRIPTION:
Improved survival after solid organ transplantation has created the need to better prevent the long-term adverse effects of immunosuppressant drugs in transplant survivors - particularly cancer development. Keratinocyte carcinoma (non-melanoma skin cancer) is by far the most common form of post-transplant malignancy and has a more aggressive clinical course than in the general population. Preventive measures are thus critical to reduce the burden of skin cancer in the high-risk transplant population.

Nicotinamide is a low-cost, commercially available, over-the-counter Vitamin B3 derivative that has been found to safely reduce the rate of keratinocyte carcinoma in immunocompetent patients with a history of skin cancer. It is unclear whether its efficacy and safety translate to the immunosuppressed transplant population.

Given this uncertainty, Investigators plan to build on our internal pilot study (N=120) to conduct the SPRINTR (Skin cancer PRevention with Nicotinamide in Transplant Recipients) pivotal trial to address these specific aims:

Primary question: Does oral nicotinamide (500 mg twice daily) reduce the rate of further keratinocyte carcinoma compared with placebo when used in addition to standard care for up to 208 weeks in high-risk solid organ transplant recipients?

Secondary questions:

1. What is the safety of nicotinamide when used in addition to standard care for up to 208 weeks in the transplant population?
2. What is the effect of nicotinamide on quality of life related to skin cancer?

Investigators will conduct a multicentre, pragmatic, parallel group, investigator- and patient-blinded, randomized trial with a superiority framework. This pivotal trial will evaluate the efficacy and safety of oral nicotinamide versus placebo to prevent further keratinocyte carcinoma in 396 high-risk solid organ transplant recipients. Data from our previous internal pilot study (N=120 participants) will be combined with data from the current pivotal trial (N=276 additional patients) in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Kidney, liver, heart, or lung transplant at least two years ago
* History of at least one prior histologically-confirmed keratinocyte carcinoma or squamous cell carcinoma in situ
* Currently immunosuppressed with a calcineurin inhibitor-based regimen (cyclosporine or tacrolimus)
* Able to attend follow-up visits

Exclusion Criteria:

* Use of nicotinamide or niacin (≥250 mg daily) within past 12 weeks
* Untreated localized skin cancer at baseline (patient can enrol after skin cancer treatment)
* Biopsy-confirmed acute rejection episode within the past 12 weeks
* Active liver disease (high AST >3 times or bilirubin >1.5 times)
* Severe kidney disease (estimated glomerular filtration rate <20 mL/min/1.73 m2)
* Solid organ or hematologic malignancy, invasive melanoma, Merkel cell carcinoma, or metastatic skin cancer within the past five years
* Pregnancy or lactation
* Need for ongoing carbamazepine or primidone
* Allergy to nicotinamide or any ingredient of the vitamin or placebo capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Time to first biopsy-confirmed keratinocyte carcinoma (basal cell carcinoma or invasive cutaneous squamous cell carcinoma) | Up to 208 weeks

SECONDARY OUTCOMES:
Time to first invasive squamous cell carcinoma during follow-up | Up to 208 weeks
Time to first basal cell carcinoma during follow-up | Up to 208 weeks
Time to multiple keratinocyte carcinomas over follow-up | Up to 208 weeks
Occurrence of adverse events during follow-up | 208 weeks
  Overall and by body system, frequency, seriousness, and severity
Acute graft rejection (biopsy-confirmed) | 208 weeks
  Adverse event
Graft loss or retransplantation | 208 weeks
  Adverse event
High/low cyclosporine or tacrolimus blood concentration requiring dose adjustment | 208 weeks
  Adverse event
Change from baseline in annual Basal and Squamous Cell Carcinoma Quality of Life (BaSQoL) score | 52 weeks
Change from baseline in annual Basal and Squamous Cell Carcinoma Quality of Life (BaSQoL) score | 104 weeks
Change from baseline in annual Basal and Squamous Cell Carcinoma Quality of Life (BaSQoL) score | 156 weeks
Change from baseline in annual Basal and Squamous Cell Carcinoma Quality of Life (BaSQoL) score | 208 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Montreal Cognitive Assessment (MoCA) | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Montreal Cognitive Assessment (MoCA) | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Montreal Cognitive Assessment (MoCA) | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Montreal Cognitive Assessment (MoCA) | 208 weeks
Neurocognitive substudy - Proportion of participants with cognitive impairment | 52 weeks
  As defined by the International Cognition and Cancer Task Force (T scores ≥2 standard deviations below the normative population mean on a single test, or ≥1.5 standard deviations below the mean on at least two tests, or both)
Neurocognitive substudy - Proportion of participants with cognitive impairment | 104 weeks
  As defined by the International Cognition and Cancer Task Force (T scores ≥2 standard deviations below the normative population mean on a single test, or ≥1.5 standard deviations below the mean on at least two tests, or both)
Neurocognitive substudy - Proportion of participants with cognitive impairment | 156 weeks
  As defined by the International Cognition and Cancer Task Force (T scores ≥2 standard deviations below the normative population mean on a single test, or ≥1.5 standard deviations below the mean on at least two tests, or both)
Neurocognitive substudy - Proportion of participants with cognitive impairment | 208 weeks
  As defined by the International Cognition and Cancer Task Force (T scores ≥2 standard deviations below the normative population mean on a single test, or ≥1.5 standard deviations below the mean on at least two tests, or both)
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Hopkins Verbal Learning Test - Revised | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Hopkins Verbal Learning Test - Revised | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Hopkins Verbal Learning Test - Revised | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Hopkins Verbal Learning Test - Revised | 208 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Trail Making A and B | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Trail Making A and B | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Trail Making A and B | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Trail Making A and B | 208 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Controlled Oral Word Association | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Controlled Oral Word Association | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Controlled Oral Word Association | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Controlled Oral Word Association | 208 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Animal Naming Task | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Animal Naming Task | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Animal Naming Task | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Animal Naming Task | 208 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Wechsler Adult Intelligence Scale-Fourth Edition-Canadian (WAIS-IV-CDN). | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Wechsler Adult Intelligence Scale-Fourth Edition-Canadian (WAIS-IV-CDN). | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Wechsler Adult Intelligence Scale-Fourth Edition-Canadian (WAIS-IV-CDN). | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Wechsler Adult Intelligence Scale-Fourth Edition-Canadian (WAIS-IV-CDN). | 208 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Digit Span subtest | 52 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Digit Span subtest | 104 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Digit Span subtest | 156 weeks
Neurocognitive substudy - Change from baseline in demographically-corrected T score for Digit Span subtest | 208 weeks

CONTACTS AND LOCATIONS:
Overall Officials: An-Wen Chan, Principal Investigator — Women's College Hospital; Sang Joseph Kim, Principal Investigator — University Health Network, Toronto
Locations (7):
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol and statistical code will be shared upon request. Beyond 18 months after trial completion, the anonymized participant-level dataset will made available for sharing with external researchers upon approval of a reasonable study proposal describing the intended data usage.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beyond 18 months after trial completion.
Access Criteria: Data will be made available for sharing with external researchers upon approval of a well-defined study proposal that clearly outlines the intended use of the data.